CLINICAL TRIAL: NCT06038383
Title: Effect of Physical Exercise Performed Through Virtual Reality Games on the Modulation of Heart Rate Variability in Chronic Renal Patients During Hemodialysis.
Brief Title: Effect of Physical Exercise Performed Through Virtual Reality Games on Chronic Renal Patients During Hemodialysis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Talita Dias da Silva-Magalhães, Researcher, University of Sao Paulo
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 5.802.024
Record Dates: First submitted 2023-08-29; First posted 2023-09-14 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Renal Insufficiency, Chronic
Keywords: hemodialysis; physical exercise; virtual reality; Renal Insufficiency; heart rate variability
MeSH Terms: conditions — Renal Insufficiency, Chronic; Motor Activity; Renal Insufficiency | interventions — Cross-Over Studies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group A - Intervention with Virtual Reality (VR) (Experimental): Group of people with kidney disease that enrolled the intervention with VR during hemodialysis.
  Interventions: Device: Group A - Intervention with Virtual Reality (VR)
- Group B - Intervention with Stationary Bike (SB) (Active Comparator): Group of people with kidney disease that enrolled the intervention with SB during hemodialysis.
  Interventions: Device: Group B - Intervention with Stationary Bike (SB)
- Group A - Intervention with Stationary Bike (SB) - Crossover (Experimental): Group of people with kidney disease that enrolled the intervention with SB during hemodialysis, after the period of washout.
  Interventions: Device: Group A - Intervention with Stationary Bike (SB) - Crossover
- Group B - Intervention with Virtual Reality (VR) - Crossover (Active Comparator): Group of people with kidney disease that enrolled the intervention with VR during hemodialysis, after the period of washout.
  Interventions: Device: Group B - Intervention with Virtual Reality (VR) - Crossover

INTERVENTIONS:
Device: Group A - Intervention with Virtual Reality (VR) — Group of people with kidney disease that performed VR intervention during hemodialysis.
  Arms: Group A - Intervention with Virtual Reality (VR)
Device: Group B - Intervention with Stationary Bike (SB) — Group of people with kidney disease that performed SB intervention during hemodialysis.
  Arms: Group B - Intervention with Stationary Bike (SB)
Device: Group A - Intervention with Stationary Bike (SB) - Crossover — Group of people with kidney disease that performed SB intervention during hemodialysis after the washout period.
  Arms: Group A - Intervention with Stationary Bike (SB) - Crossover
Device: Group B - Intervention with Virtual Reality (VR) - Crossover — Group of people with kidney disease that performed VR intervention during hemodialysis after the washout period.
  Arms: Group B - Intervention with Virtual Reality (VR) - Crossover

SUMMARY:
Patients with chronic kidney diseases, especially those requiring hemodialysis, are characterized by an increased risk of numerous morbidities. This is a condition that significantly impacts the patient's quality of life, leads to dependence, and involves high-cost treatment. The physical condition of chronic kidney disease patients falls well below the recommendations set by the World Health Organization, indicating effective difficulties in the approaches used for implementing physical activity programs. New approaches must be considered. Physical activity through virtual reality can foster greater social integration of patients with physical exercise during hemodialysis, enabling improved quality of life and decreased frailty levels for these individuals due to its playful and motivational nature.

Objective: To assess changes in heart rate variability modulation and the quality of life of chronic kidney disease patients undergoing virtual reality-based exercise during hemodialysis sessions.

Methods: A longitudinal, controlled, randomized crossover clinical trial. The chronic kidney disease groups will be divided into two groups, Group A (GA) and Group B (GB). Group GA will engage in 10 interventions, with each intervention involving the completion of 3 sessions of a Virtual Reality (VR) game lasting 5 minutes each, totaling 15 minutes of exercise. Group GB will participate in 10 interventions, with each intervention comprising 15 minutes of physical exercise on a cycle ergometer, referred to here as conventional exercise.

After the initial 10 interventions, the groups will switch exercises; that is, GA will cease VR interventions and begin another 10 interventions with conventional exercise, while GB will stop conventional exercise interventions and start another 10 interventions with VR.

The Kidney Disease Quality of Life Short Form questionnaire, Beck's Anxiety and Depression Inventory, and the International Physical Activity Questionnaire will also be administered to all groups.

DETAILED DESCRIPTION:
The objective of this Longitudinal CrossOver Clinical Trial is to compare changes in heart rate variability modulation in chronic renal patients undergoing conventional physical exercise and in a virtual environment during hemodialysis sessions.

The main questions it aims to answer are:

What are the differences in changes in heart rate variability modulation between chronic renal patients who undergo conventional physical exercise before and during hemodialysis sessions, and those who engage in virtual environment exercises?

How does the virtual environment influence changes in heart rate variability modulation compared to conventional physical exercise in chronic renal patients before and during hemodialysis sessions?

What is the relative effectiveness of conventional physical exercise compared to virtual environment exercise in improving heart rate variability modulation in chronic renal patients before and during hemodialysis sessions?

Group A will participate in 10 interventions, each intervention consisting of playing 3 rounds of a Virtual Reality game lasting 5 minutes, totaling 15 minutes of exercise. Group B will participate in 10 interventions, each intervention consisting of 15 minutes of physical exercise on a cycle ergometer, referred to here as conventional exercise.

After the initial 10 interventions,there will be a 1-week washout period and the groups will switch exercises. Heart rate and respiratory rate, oxygen saturation, systemic blood pressure, laboratory tests, as well as the Kidney Disease Quality of Life Short Form questionnaire, the Beck Anxiety and Depression Inventory, and the International Physical Activity Questionnaire will be assessed in all groups.

ELIGIBILITY:
Inclusion Criteria:

* Patients with diagnosed chronic renal insufficiency requiring hemodialysis at any classification level.
* Age over 18 years.
* Possession of medical clearance for participating in physical exercise.
* Ability for lower limb movement without affecting dialysis treatment.

Exclusion Criteria:

* Acute use of medications that affect the cardiovascular system and/or alter the function of the nervous system, unless they are part of the disease treatment protocol and are part of the patient's routine.
* Reports of persistent pain and fatigue arising after the start of exercise training.
* Changes in the type of renal treatment during the protocol application period.
* Absence from three consecutive exercise training sessions.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
Heart Rate Variability behavior during interventions with Virtual Reality and Stationary Bike while in hemodialysis. | 4 days
  Measurements made by heart rate variability indices, using both linear and non-linear measurements, using a chest trap that captures the R-R intervals in milliseconds.

SECONDARY OUTCOMES:
Blood pressure during interventions with Virtual Reality and Stationary Bike while in hemodialysis | 20 days
  Measurements made by blood pressure in mmHg
Heart rate during interventions with Virtual Reality and Stationary Bike while in hemodialysis | 20 days
  Measurements made by heart rate in beats per minute.
Respiratory rate during interventions with Virtual Reality and Stationary Bike while in hemodialysis | 20 days
  Measurements made by respiratory rate in incursions per minute.
Oxygen saturation during interventions with Virtual Reality and Stationary Bike while in hemodialysis | 20 days
  Measurements made by oxygen saturation in percentage.

CONTACTS AND LOCATIONS:
Overall Officials: Talita D Silva, PhD, Principal Investigator — Federal University of São Paulo
Locations (1):
- Comitê de Etica da Universidade Federal de São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No